CLINICAL TRIAL: NCT03265288
Title: APPLAUD: A Double-Blind, Randomized, Placebo-Controlled, Phase II Study of the Efficacy and Safety of LAU-7b in the Treatment of Cystic Fibrosis in Adults
Brief Title: Study of LAU-7b in the Treatment of Cystic Fibrosis in Adults
Acronym: APPLAUD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Laurent Pharmaceuticals Inc. (Industry)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LAU-14-01
Record Dates: First submitted 2017-02-21; First posted 2017-08-29 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Cystic Fibrosis
Keywords: Inflammation; Essential Fatty Acids; Inflammation resolution; Docosahexaenoic acid; Lung function
MeSH Terms: conditions — Cystic Fibrosis; Inflammation | interventions — Fenretinide

STUDY DESIGN:
Intervention Model Description: Double-blind, randomized, parallel groups and placebo-controlled trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Patients will be randomly assigned to take either the active drug (fenretinide capsule) or a matching inactive placebo (inactive capsule).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- LAU-7b (Experimental): Active drug fenretinide (as LAU-7b capsules)
  Interventions: Drug: LAU-7b
- Placebo (Placebo Comparator): Placebo oral capsule (as inactive capsules identical to active arm)
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: LAU-7b — LAU-7b will be administered orally once-a-day with the first meal of the day as cycles of 21 days on, 7 days off, for a total of 6 planned cycles.
  Other Names: fenretinide
  Arms: LAU-7b
Drug: Placebo oral capsule — Placebo will be administered orally once-a-day with the first meal of the day as cycles of 21 days on, 7 days off, for a total of 6 planned cycles.
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
An International Phase II, double-blind, randomized, placebo-controlled study to evaluate the safety and efficacy of LAU-7b administered once-daily for 6 months for the treatment of CF.

DETAILED DESCRIPTION:
An International Phase II, double-blind, randomized, placebo-controlled study to evaluate the safety and efficacy of LAU-7b administered once-daily for 6 months for the treatment of CF. All patients will remain on their CF standard-of-care treatments over the trial duration.

The goal for the treatment with LAU-7b in CF is to preserve lung function by reducing the persistent inflammation in the lung and to improve its capacity to defend against resistant bacteria such as Pseudomonas aeruginosa.

The treatment regimen will consist of 6 consecutive "dosing cycles" of 21 days each, spaced by study drug-free periods of 7 days. A total of 136 eligible adult patients with CF will be randomized to receive 300 mg LAU-7b or placebo in a 1:1 ratio. The participation in the study will last about 7 months.

ELIGIBILITY:
Inclusion Criteria:

* Screening FEV1 between 40% and 100% predicted value for age, gender and height, in patients capable of properly performing the test;
* History of pulmonary exacerbation, defined as at least one (1) pulmonary exacerbation in the year prior to Screening which resulted in documented intravenous or Oral antibiotics;
* Patients are eligible independently of their history of pulmonary Pseudomonas aeruginosa (PsA) infection and their PsA status at screening;
* If taking Kalydeco® (ivacaftor), Orkambi® (ivacaftor/lumacaftor), Symdeko® (ivacaftor/tezacaftor) or other commercially available CFTR modulator products, patients must be taking it for a minimum of 3 months prior to screening if naïve to CFTR modulators and 1 month if switched from another CFTR modulator product and deemed to tolerate it;
* No change in CF and allowed systemic chronic therapy for a minimum of 5 weeks prior to randomization, of which 2 weeks minimum are prior to screening;
* Female patients of child bearing potential should be on highly effective contraceptive methods during the study;
* Male patients with spouse or partner of child bearing potential, or pregnant, are eligible if they use an appropriate method of contraception.

Exclusion Criteria:

* Pregnancy: due to the potential teratogenic effects of retinoids, pregnant women are NOT eligible;
* Breast milk feeding by study patient is NOT allowed;
* Clinically abnormal renal function: serum creatinine > 132 μM (1.5 mg/dL);
* Clinically abnormal liver function: Total bilirubin >1.5 x ULN (in the absence of demonstrated Gilbert's syndrome), alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 2.5 x ULN;
* Patients with plasma retinol levels below 0.7 µM;
* Presence of nyctalopia or hemeralopia at enrolment, or any other serious retinal, ophthalmological condition;
* Presence of serious dermatological conditions at entry, including inflammatory or xerotic skin pathologies such as psoriasis or ichthyosis;
* Intake of chronic systemic steroids in the month prior to screening and during the study;
* History of acute infections (viral/bacterial/fungal) within 5 weeks prior to randomization, of which 2 weeks minimum are prior to screening, whether or not treated and resolved;
* Presence of infection with Burkholderia cepacia (including all species within the Burkholderia cepacia complex group, and Burkholderia gladioli) in the 12 months prior to screening;
* Patients with a confirmed diagnosis (as per the Cystic Fibrosis Foundation diagnostic criteria) of Allergic BronchoPulmonary Aspergillosis (ABPA) and actively being treated with corticosteroids and/or anti fungal agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2018-11-05 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry C Lands, MD PhD, Study Chair — McGill Uinversity Health Centre; Michael W Konstan, MD, Study Chair — Rainbow Babies and Children's Hospital/ University Hospitals Cleveland Medical Center
Locations (40):
- United States (27):
  - Long Beach Memorial Medical Center, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - UC Davis Medical Center, Division of Pulmonary & Critical Care Medicine, Sacramento, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Division of pulmonary, critical care and sleep medicine, University of Florida, Gainesville, Florida
  - Memorial Healthcare System, Joe DiMaggio Children's Hospital Cystic Fibrosis & Pulmonary Center, Hollywood, Florida
  - Avanza Medical Research Center, Pensacola, Florida
  - St-Luke's CF Center of Idaho, Boise, Idaho
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Maine Medical Center Cystic Fibrosis Research, Portland, Maine
  - University of Michigan Health System, Ann Arbor, Michigan
  - Wayne State University, Harper University Hospital, Detroit, Michigan
  - The Minnesota Cystic Fibrosis Center, University of Minnesota, Minneapolis, Minnesota
  - Washington University Medical School, St Louis, Missouri
  - Morristown Medical Center, NJ Adult Cystic Fibrosis Center, Morristown, New Jersey
  - Rutgers University Clinical Research Center, RW Johnson University Hospital, New Brunswick, New Jersey
  - Albany Medical College, Albany, New York
  - University Hospitals Cleveland Medical Center, Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Cystic Fibrosis Center, Doernbecher Children's Hospital, Oregon Health & Science University, Portland, Oregon
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - Medical College of Wisconsin, Div of Pulmonary and Critical Care Medicine, Milwaukee, Wisconsin
- Australia (7):
  - Respiratory Medicine, John Hunter Hospital, New Lambton Heights, New South Wales
  - Department of Respiratory Medicine, Royal Prince Alfred Hospital, Sydney, New South Wales
  - Department of Respiratory and Sleep Medicine, Westmead Hospital, Westmead, New South Wales
  - Mater Misericordiae Ltd, Brisbane, Queensland
  - Monash Lung and Sleep, Monash Health, Clayton, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Institute of Respiratory Health, Harry Perkins Institute, Nedlands, Western Australia
- Canada (6):
  - Pacific Lung Research Institute at St. Paul's Hospital, Vancouver, British Columbia
  - The Ottawa Hospital Center for Practice-Changing Research, Ottawa, Ontario
  - Centre d'études cliniques CIUSS SLJ, Hôpital Chicoutimi, Chicoutimi, Quebec
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec
  - McGill University Health Center, Montreal, Quebec
  - Centre de recherche de l'institut Universitaire de Cardiologie et de Pneumologie de Québec, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LAU-7b | Placebo
Started | 83 | 83
Completed | 60 | 71
Not Completed | 23 | 12
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 13 | 5
Not completed — Drug Withdrawn | 3 | 3
Not completed — Any Other Reason | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LAU-7b | Placebo | Total
Number analyzed (Participants) | 83 | 83 | 166
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.5 (10.70) | 33.9 (12.95) | 32.7 (11.90)
Age, Customized [Count of Participants; unit: Participants]
  <=25 years | 29 | 26 | 55
  >25 years | 54 | 57 | 111
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 49 | 99
  Male | 33 | 34 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 2 | 9
  Not Hispanic or Latino | 76 | 81 | 157
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 81 | 78 | 159
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 24 | 22 | 46
  United States | 48 | 51 | 99
  Australia | 11 | 10 | 21
Weight (kg), Mean (SD) [Mean (Standard Deviation); unit: kg] | 63.88 (12.213) | 64.53 (14.329) | 64.20 (13.277)
BMI (kg/m2), Mean (SD) [Mean (Standard Deviation); unit: kg/m2] | 23.34 (3.354) | 23.39 (4.099) | 23.36 (3.734)
Number of PEx in the previous year, (Mean (SD) [Mean (Standard Deviation); unit: Pulmonary Exacerbation] | 2.3 (1.77) | 2.1 (1.54) | 2.2 (1.65)
FEV1 percent predicted at Baseline [Mean (Standard Deviation); unit: percent predicted] | 63.2 (16.77) | 62.3 (15.13) | 62.73 (15.93)

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Percent Predicted Forced Expiratory Volume in 1 Second (FEV1%)
Description: Standardized, serial FEV1 measurements were performed during the trial by the clinical sites using standardized spirometers. All spirometry measurements were centrally read and validated by the spirometry provider, Vitalograph. The outcome measure is presented using the Least Squares Mean at the Week 24 time point and the Least Squares Mean of all post-baseline time points through Week 24 averaged.
Time Frame: From baseline to 24 weeks
Population: intent to treat population (ITT) and per-protocol population (PP)
Measure: Least Squares Mean (95% Confidence Interval); unit: Change in FEV1 % predicted
Groups:
- LAU-7b: Active drug fenretinide (as LAU-7b capsules)
  LAU-7b: LAU-7b administered orally once-a-day as cycles of 21 days on, 7 days off, for a total of 6 planned cycles.
- Placebo: Placebo oral capsule (as inactive capsules identical to active arm)
  Placebo oral capsule: Placebo administered orally once-a-day as cycles of 21 days on, 7 days off, for a total of 6 planned cycles.
Arm/Group | LAU-7b | Placebo
Number analyzed (Participants) | 83 | 83
Change in FEV1 % predicted
  ITT population at Week 24 | -1.1774 [-2.5038 to 0.1490] | -1.9489 [-3.2241 to -0.6738]
  ITT population through Week 24 | -0.5417 [-1.5226 to 0.4392] | -1.5470 [-2.5304 to -0.5637]
  PP population through Week 24: number analyzed (Participants) | 55 | 67
  PP population through Week 24 | -0.3374 [-1.4987 to 0.8239] | -1.5632 [-2.7333 to -0.3930]
  ITT subgroup >=70% ppFEV1, at Week 24: number analyzed (Participants) | 29 | 27
  ITT subgroup >=70% ppFEV1, at Week 24 | -1.4059 [-3.5506 to 0.7388] | -4.0687 [-6.1289 to -2.0085]
  ITT subgroup on CFTR modulators, at Week 24: number analyzed (Participants) | 41 | 46
  ITT subgroup on CFTR modulators, at Week 24 | -0.3336 [-2.2467 to 1.5795] | -1.7247 [-3.2954 to -0.1539]
  ITT subgroup on ETI, at Week 24: number analyzed (Participants) | 18 | 23
  ITT subgroup on ETI, at Week 24 | -0.7406 [-3.7472 to 2.2659] | -1.8709 [-4.1669 to 0.4252]
Statistical Analysis 1: Comparison: LAU-7b vs Placebo; Primary analysis of the treatment effect at the Week 24 visit on the intent to treat population (ITT) Null hypothesis is no treatment difference; Test type: Superiority; p = 0.3449, Mixed Model for Repeated Measures — alpha is set to 0.05; Least square means difference = 0.7716, 95% CI 2-sided [-0.8397 to 2.3828] — A positive difference favours LAU-7b, a negative difference favours placebo
Statistical Analysis 2: Comparison: LAU-7b vs Placebo; Analysis of the overall treatment effect from baseline through Week 24 in the intent to treat population (ITT), Null hypothesis is no treatment difference; Test type: Superiority; p = 0.0667, Mixed Model for Repeated Measures — alpha is set to 0.05; Least square means difference = 1.0053, 95% CI 2-sided [-0.0700 to 2.0807] — A positive difference favours LAU-7b, a negative difference favours placebo
Statistical Analysis 3: Comparison: LAU-7b vs Placebo; Secondary analysis of the overall treatment effect from baseline through Week 24 on the per protocol population (PP), null hypothesis is no treatment difference; Test type: Superiority; p = 0.0486, Mixed Model for Repeated Measures — alpha is set to 0.05; Least square means difference = 1.2258, 95% CI 2-sided [0.0078 to 2.4438] — A positive difference favours LAU-7b, a negative difference favours placebo
Statistical Analysis 4: Comparison: LAU-7b vs Placebo; Secondary analysis of treatment effect at the Week 24 visit for stratification factor ppFEV1 (<70% or ≥70%) in intent to treat population (ITT), null hypothesis is no treatment difference. Here presented is the analysis for subgroup ≥70%, n=29 (LAU-7b), n=27 (Placebo); Test type: Superiority; p = 0.0687, Mixed Model for Repeated Measures — alpha is set to 0.05; Least square means difference = 2.6628, 95% CI 2-sided [-0.2069 to 5.5325] — A positive difference favours LAU-7b, a negative difference favours placebo
Statistical Analysis 5: Comparison: LAU-7b vs Placebo; Secondary analysis of treatment effect at the Week 24 visit for stratification factor co-administration of CFTR modulator (yes/no) in intent to treat population (ITT), null hypothesis is no treatment difference. Here presented is the analysis for subgroup receiving CFTR modulators, n=41 (LAU-7b), n=46 (Placebo); Test type: Superiority; p = 0.236, Mixed Model for Repeated Measures — alpha is set to 0.05; Least square means difference = 1.391, 95% CI 2-sided [-0.9220 to 3.7041] — A positive difference favours LAU-7b, a negative difference favours placebo
Statistical Analysis 6: Comparison: LAU-7b vs Placebo; Secondary analysis of treatment effect at the Week 24 visit for à priori defined subgroup co-administration of ETI - elexacaftor/tezacaftor/ivacaftor (yes/no) in intent to treat population (ITT), null hypothesis is no treatment difference. Here presented is the analysis for subgroup receiving ETI, n=18 (LAU-7b), n=23 (Placebo); Test type: Superiority; p = 0.5323, Mixed Model for Repeated Measures — alpha is set to 0.05; Least square means difference = 1.1302, 95% CI 2-sided [-2.4447 to 4.7052] — A positive difference favours LAU-7b, a negative difference favours placebo

2. Primary Outcome: Summary of Treatment Emergent Adverse Events With ≥ 10% Incidence
Description: This was assessed through adverse event monitoring at all visits, including spontaneously reported events and those obtained through serial probing of the subjects, and from safety laboratory tests
Time Frame: From Baseline to 28 weeks
Population: safety population
Measure: Count of Participants; unit: Participants
Arm/Group | LAU-7b | Placebo
Number analyzed (Participants) | 83 | 83
Participants
  Subjects with at least one TEAE with ≥10% incidence | 74 | 64
  Mild highest reported severity | 22 | 27
  Moderate highest reported severity | 45 | 43
  Severe highest reported severity | 13 | 7
  Life threatening | 0 | 0
  Infective pulmonary exacerbation of cystic fibrosis | 37 | 32
  Cough | 23 | 24
  Delayed dark adaptation | 22 | 4
  Night blindness | 15 | 2
  Headache | 14 | 10
  Upper respiratory tract infections | 13 | 8
  Hemoptysis | 11 | 13
  Diarrhoea | 11 | 6
  Fatigue | 10 | 7
  Delayed light adaptation | 10 | 2
  Dyspnea | 10 | 11
  Glare | 9 | 6
  Visual impairment | 9 | 2
  Sputum increased | 7 | 13

3. Secondary Outcome: The Proportion of Patients Achieving Normalization of the Arachidonic Acid, Docosahexaenoic Acid and Their Ratio in Phospholipids
Description: Assessed through 4 blood sampling occasions during the trial. Plasma samples were analyzed using a validated LC/MS method and corrected for phospholipid content. Highest proportion of normalization during treatment was determined versus analyte ranges obtained from a group of 20 healthy, non-CF individuals.
Time Frame: From baseline to 28 weeks
Population: Intent to treat population with analytical results at any sampling visit up to 28 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | LAU-7b | Placebo
Number analyzed (Participants) | 58 | 61
Participants
  Arachidonic acid (AA) normalization | 15 | 25
  Docosahexaenoic acid (DHA) normalization | 16 | 18
  AA/DHA ratio normalization | 25 | 23
Statistical Analysis 1: Comparison: LAU-7b vs Placebo; Highest normalization of Arachidonic Acid (AA) during treatment Intent to treat population (ITT), null hypothesis is no treatment effect; Test type: Superiority; p = 0.1047, Regression, Logistic — alpha is set to 0.05; Odds Ratio (OR) = 0.5036, 95% CI 2-sided [0.2199 to 1.1532] — Odds ratio < 1 means lower odds of normalization with LAU-7b, odds ratio > 1 means higher odds of normalization with LAU-7b
Statistical Analysis 2: Comparison: LAU-7b vs Placebo; Highest normalization of Docosahexaenoic Acid (DHA) during treatment Intent to treat population (ITT, null hypothesis is no treatment effect; Test type: Superiority; p = 0.7596, Regression, Logistic — alpha is set to 0.05; Odds Ratio (OR) = 0.8773, 95% CI 2-sided [0.3793 to 2.0291] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: LAU-7b vs Placebo; Highest normalization of AA/DHA ratio during treatment Intent to treat population (ITT), null hypothesis is no treatment effect; Test type: Superiority; p = 0.8852, Regression, Logistic — alpha is set to 0.05; Odds Ratio (OR) = 1.0532, 95% CI 2-sided [0.5209 to 2.1296] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: The Absolute Change in FEV1 Percent Predicted at 3, 7, 11, 15, 24 and 28 Weeks Into the Trial
Description: Standardized, serial FEV1 measurements were performed during the trial by the clinical sites using standardized spirometers. All spirometry measurements were centrally read and validated by the spirometry provider, Vitalograph.
Time Frame: From baseline to 3, 7, 11, 15, 24 and 28 weeks into the trial
Population: Intent to treat population (ITT)
Measure: Mean (Standard Deviation); unit: FEV1 percent predicted change
Arm/Group | LAU-7b | Placebo
Number analyzed (Participants) | 83 | 83
FEV1 percent predicted change
  Absolute change at Week 3 | -0.243 (5.110) | -1.494 (4.537)
  Absolute change at Week 7 | 0.280 (4.689) | -0.888 (3.968)
  Absolute change at Week 11 | -0.309 (4.268) | -0.871 (4.133)
  Absolute change at Week 15 | -0.508 (5.100) | -1.591 (4.389)
  Absolute change at Week 24 | -1.024 (4.286) | -1.759 (4.533)
  Absolute change at Week 28 | -1.539 (4.808) | -1.413 (4.457)

5. Secondary Outcome: The Relative (%) Change in FEV1 Percent Predicted at 3, 7, 11, 15, 24 and 28 Weeks Into the Trial
Description: as for outcome 4
Time Frame: From baseline to 3, 7, 11, 15, 24 and 28 weeks into the trial
Population: Intent to treat population (ITT)
Measure: Mean (Standard Deviation); unit: FEV1 percent predicted change
Arm/Group | LAU-7b | Placebo
Number analyzed (Participants) | 83 | 83
FEV1 percent predicted change
  Relative (%) change at Week 3 | -1.188 (8.632) | -2.341 (7.289)
  Relative (%) change at Week 7 | 0.561 (8.348) | -1.550 (6.829)
  Relative (%) change at Week 11 | -0.213 (7.124) | -1.277 (7.120)
  Relative (%) change at Week 15 | -0.924 (8.963) | -2.745 (7.425)
  Relative (%) change at Week 24 | -1.450 (6.966) | -2.652 (7.742)
  Relative (%) change at Week 28 | -2.388 (8.275) | -2.085 (7.525)

6. Secondary Outcome: The Time to First Protocol-Defined Pulmonary Exacerbation
Description: Reports of IV antibiotics-treated pulmonary exacerbations during the trial that meet the Fuch's criteria and after the first treatment cycle.
Time Frame: From baseline to 28 weeks
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | LAU-7b | Placebo
Number analyzed (Participants) | 83 | 83
days | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events
Statistical Analysis 1: Comparison: LAU-7b vs Placebo; Test type: Superiority; p = 0.3025, Log Rank

7. Secondary Outcome: The Number Per Subject of Protocol-Defined Pulmonary Exacerbations (PEx) During the Trial
Description: The number per subject of Protocol-Defined IV antibiotics-treated pulmonary exacerbations (events) during the trial that meet the Fuch's criteria. Also presented are the number per subject of IV antibiotics-treated pulmonary exacerbations and combined number per subject of IV- or Oral antibiotics-treated pulmonary exacerbations during the trial. Excluded are exacerbations occurring during the first treatment cycle.
Time Frame: From baseline to 28 weeks
Measure: Mean (Standard Deviation); unit: Events per subject
Arm/Group | LAU-7b | Placebo
Number analyzed (Participants) | 83 | 83
Events per subject
  Protocol-Defined IV-treated PEx events per subject | 0.16 (0.398) | 0.10 (0.335)
  All IV-treated PEx events per subject | 0.24 (0.458) | 0.18 (0.566)
  All IV- or Oral antibiotics-treated PEx events per subject | 0.53 (0.721) | 0.47 (0.817)
Statistical Analysis 1: Comparison: LAU-7b vs Placebo; Protocol-Defined IV antibiotics-treated pulmonary exacerbation events. Intent to treat population (ITT), null hypothesis is no treatment effect; Test type: Superiority; p = 0.3366, Regression, Cox — alpha is set to 0.05; Risk Ratio (RR) = 1.55, 95% CI 2-sided [0.63 to 3.80] — Odds ratio < 1 means lower odds of a pulmonary exacerbation with LAU-7b, odds ratio close to 1 means similar odds of a pulmonary exacerbation for LAU-7b and placebo, odds ratio > 1 means higher odds of a pulmonary exacerbation with LAU-7b
Statistical Analysis 2: Comparison: LAU-7b vs Placebo; ALL IV antibiotics-treated pulmonary exacerbation events. Intent to treat population (ITT), null hypothesis is no treatment effect; Test type: Other; p = 0.3936, Regression, Cox — alpha is set to 0.05; Risk Ratio (RR) = 1.34, 95% CI 2-sided [0.68 to 2.64] — [estimate comment as in outcome 7, analysis 1]
Statistical Analysis 3: Comparison: LAU-7b vs Placebo; Combined IV- or Oral antibiotics-treated pulmonary exacerbation events. Intent to treat population (ITT), null hypothesis is no treatment effect; Test type: Superiority; p = 0.5011, Regression, Cox — alpha is set to 0.05; Risk Ratio (RR) = 1.16, 95% CI 2-sided [0.75 to 1.79] — [estimate comment as in outcome 7, analysis 1]

8. Secondary Outcome: The Time to First Change and Usage of Antibiotic (Other Than Chronic Inhaled Antibiotics Already Started Prior to Trial or Oral Chronic Azithromycin)
Description: The time to first change and usage of IV antibiotics to treat pulmonary exacerbations during the trial. Excluded are exacerbations occurring during the first treatment cycle.
Time Frame: From baseline to 28 weeks
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | LAU-7b | Placebo
Number analyzed (Participants) | 83 | 83
days | NA [NA to NA] — Insufficient number of participants with events | NA [NA to NA] — Insufficient number of participants with events
Statistical Analysis 1: Comparison: LAU-7b vs Placebo; Test type: Superiority; p = 0.1955, Log Rank

9. Secondary Outcome: Usage (Number of Antibiotic Treatments) of Antibiotic (Other Than Chronic Inhaled Antibiotics Already Started Prior to Trial or Oral Chronic Azithromycin)
Description: Usage (number of antibiotic treatments per subject) of IV antibiotics to treat pulmonary exacerbations during the trial. Excluded are exacerbations occurring during the first treatment cycle.
Time Frame: From baseline to 28 weeks
Measure: Mean (Standard Deviation); unit: Number of IV antibiotic treatments
Arm/Group | LAU-7b | Placebo
Number analyzed (Participants) | 83 | 83
Number of IV antibiotic treatments | 0.53 (1.09) | 0.41 (1.32)
Statistical Analysis 1: Comparison: LAU-7b vs Placebo; Number per subject of intravenous antibiotic treatments required for a pulmonary exacerbation, excludes Cycle 1 pulmonary exacerbations Intent to treat population (ITT), null hypothesis is no treatment effect; Test type: Superiority; p = 0.1909, Poisson regression — alpha is set to 0.05; Risk Ratio (RR) = 1.35, 95% CI 2-sided [0.86 to 2.12] — Odds ratio < 1 means lower odds of an antibiotic treatment with LAU-7b, odds ratio > 1 means higher odds of an antibiotic treatment with LAU-7b

10. Secondary Outcome: Usage (Days) of Antibiotic (Other Than Chronic Inhaled Antibiotics Already Started Prior to Trial or Oral Chronic Azithromycin)
Description: Usage (days) of IV antibiotics to treat pulmonary exacerbations during the trial. Excluded are exacerbations occurring during the first treatment cycle.
Time Frame: From baseline to 28 weeks
Measure: Mean (Standard Deviation); unit: Days of IV antibiotics
Arm/Group | LAU-7b | Placebo
Number analyzed (Participants) | 83 | 83
Days of IV antibiotics | 3.8 (7.50) | 3.5 (14.94)
Statistical Analysis 1: Comparison: LAU-7b vs Placebo; Number of days of intravenous antibiotics required for a pulmonary exacerbation, excludes Cycle 1 pulmonary exacerbations, Intent to treat population (ITT), null hypothesis is no treatment effect; Test type: Superiority; p = 0.7473, Poisson regression — alpha is set to 0.05; Risk Ratio (RR) = 1.11, 95% CI 2-sided [0.60 to 2.04] — Odds ratio < 1 means lower odds in terms of days of antibiotics with LAU-7b, odds ratio close to 1 means similar odds in terms of days of antibiotics with LAU-7b or placebo, odds ratio > 1 means higher odds in terms of days of antibiotics with LAU-7b

11. Secondary Outcome: The Change From Baseline of Systemic Markers of Inflammation in Blood
Description: This was assessed through scheduled blood sampling during the trial on three occasions. Both ITT and PP populations results presented. Samples were analyzed using validated analytical methods.
Time Frame: Change from baseline to Week 24
Population: Intent to treat population (ITT) and per-protocol population (PP)
Measure: Mean (Standard Deviation); unit: Change in mg/L
Arm/Group | LAU-7b | Placebo
Number analyzed (Participants) | 83 | 83
Change in mg/L
  Absolute change from baseline of C-reactive protein at Week 24 ITT Population | -1.197 (7.904) | 2.532 (10.650)
  Absolute change from baseline of calprotectin at Week 24, ITT population | -27 (962) | 478 (2088)
  Absolute change from baseline of C-reactive protein at Week 24 PP Population: number analyzed (Participants) | 55 | 67
  Absolute change from baseline of C-reactive protein at Week 24 PP Population | -1.216 (7.987) | 2.532 (10.654)
  Absolute change from baseline of calprotectin at Week 24, PP population: number analyzed (Participants) | 55 | 67
  Absolute change from baseline of calprotectin at Week 24, PP population | -18 (970) | 478 (2088)
Statistical Analysis 1: Comparison: LAU-7b vs Placebo; C-Reactive Protein (CRP), Intent-to-Treat population (ITT), null hypothesis is no treatment effect; Test type: Superiority; p = 0.0822, Mixed Model for Repeated Measures — alpha is set to 0.05; Least Squares Means difference = -2.890, 95% CI 2-sided [-6.154 to 0.374] — A negative difference favours LAU-7b, a positive difference favours placebo
Statistical Analysis 2: Comparison: LAU-7b vs Placebo; Calprotectin, Intent-to-Treat population (ITT), null hypothesis is no treatment effect; Test type: Superiority; p = 0.0603, Mixed Model for Repeated Measures — alpha is set to 0.05; Least Squares Means difference = -576, 95% CI 2-sided [-1177 to 25.4] — A negative difference favours LAU-7b, a positive difference favours placebo
Statistical Analysis 3: Comparison: LAU-7b vs Placebo; C-Reactive Protein (CRP), Per-Protocol population (PP), null hypothesis is no treatment effect; Test type: Superiority; p = 0.0287, Mixed Model for Repeated Measures — alpha is set to 0.05; Least Square Means difference = -3.853, 95% CI 2-sided [-7.297 to -0.408] — A negative difference favours LAU-7b, a positive difference favours placebo
Statistical Analysis 4: Comparison: LAU-7b vs Placebo; Calprotectin, Per-Protocol population (PP), null hypothesis is no treatment effect; Test type: Superiority; p = 0.0459, Mixed Model for Repeated Measures — alpha is set to 0.05; Least Square Means difference = -620, 95% CI 2-sided [-1228 to 12] — A negative difference favours LAU-7b, a positive difference favours placebo

12. Secondary Outcome: The Change From Screening of the Body Weight
Description: This was assessed through serial weighing during the trial. Measurements performed at clinical sites using calibrated balances.
Time Frame: From screening to 28 weeks
Measure: Mean (Standard Deviation); unit: Change in kg
Arm/Group | LAU-7b | Placebo
Number analyzed (Participants) | 83 | 83
Change in kg | -0.43 (2.41) | 0.14 (1.96)
Statistical Analysis 1: Comparison: LAU-7b vs Placebo; Body weight, Intent to treat population (ITT), null hypothesis is no treatment effect; Test type: Superiority; p = 0.1006, Mixed Model for Repeated Measures — alpha is set to 0.05; Least Squares Means difference = -0.39, 95% CI 2-sided [-0.86 to 0.08]

13. Secondary Outcome: The Change From Screening of the Body Mass Index (BMI)
Description: This was assessed through serial weighing during the trial and calculation of BMI. Measurements performed at clinical sites using calibrated balances.
Time Frame: From screening to 28 weeks
Population: Intent to treat (ITT)
Measure: Mean (Standard Deviation); unit: Change in kg/m2
Arm/Group | LAU-7b | Placebo
Number analyzed (Participants) | 83 | 83
Change in kg/m2 | -0.162 (0.922) | 0.037 (0.706)
Statistical Analysis 1: Comparison: LAU-7b vs Placebo; Body mass index, intent to treat population (ITT), null hypothesis is no treatment effect; Test type: Superiority; p = 0.1246, Mixed Model for Repeated Measures — alpha is set to 0.05; Least Squares Means difference = -0.137, 95% CI 2-sided [-0.312 to 0.038]

14. Secondary Outcome: The Overall Change From Screening of the Pseudomonas Aeruginosa Density (Colony Forming Units) in the Sputum
Description: This was assessed through induced sputum (and spontaneously obtained during COVID-19 pandemic) on 3 occasions during the trial. Samples were analyzed at a central laboratory. An area under the curve (AUC from baseline to Week 24 inclusive) of colony forming unit/mL is calculated.
Time Frame: From screening to Week 24
Population: Intent to treat population (ITT) with samples at screening and post-screening timepoints, and at sites able to obtain sputum samples
Measure: Mean (Standard Deviation); unit: CFU*weeks/mL
Arm/Group | LAU-7b | Placebo
Number analyzed (Participants) | 26 | 31
CFU*weeks/mL | 17681448107 (33050105775) | 10218800226 (16808101968)
Statistical Analysis 1: Comparison: LAU-7b vs Placebo; Intent to treat population (ITT), null hypothesis is no treatment effect; Test type: Superiority; p = 0.7640, ANOVA — alpha is set to 0.05

15. Secondary Outcome: The Impact (From Baseline) on Overall Health, Daily Life, Perceived Well-being and Symptoms Measured With the Cystic Fibrosis Questionnaire-Revised (CFQ-R)
Description: This was assessed through administration of the Cystic Fibrosis Questionnaire-Revised (CFQ-R) at four planned times during the trial. The CFQ-R respiratory sub-score (range 0-100) was extracted and analyzed. The Minimum Clinically Important Difference (MCID) for the respiratory sub-score is 4 units. A higher score means a better outcome.
Time Frame: From baseline to 24 weeks
Population: Absolute change of CFQ-R Respiratory sub-score, from Baseline to Week 24. Intent to treat population (ITT)
Measure: Mean (Standard Deviation); unit: Change of units on a scale
Arm/Group | LAU-7b | Placebo
Number analyzed (Participants) | 83 | 83
Change of units on a scale | -2.485 (20.28) | 0.235 (11.44)
Statistical Analysis 1: Comparison: LAU-7b vs Placebo; CFQ-R Respiratory subscore, intent to treat population (ITT), null hypothesis is no treatment effect; Test type: Superiority; p = 0.2996, Mixed Model for Repeated Measures — alpha is set to 0.05; Least Squares Means difference = -2.758, 95% CI 2-sided [-7.998 to 2.482]

16. Secondary Outcome: The Change in Metabolipidomic Profile and in Markers of Oxidative Stress in Blood
Description: This was assessed through serial blood sampling during the trial. Samples were analyzed using validated methods at specialized laboratories.
Time Frame: From baseline to 24 weeks
Population: Absolute change from Baseline at Week 24. Intent to treat population (ITT) in subjects with samples analyzed at baseline and at Week 24
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | LAU-7b | Placebo
Number analyzed (Participants) | 83 | 83
umol/L
  11-Hydroxy Eicosatetraenoic Acid: number analyzed (Participants) | 35 | 35
  11-Hydroxy Eicosatetraenoic Acid | -0.0195 (0.13559) | 0.0187 (0.08397)
  12-Hydroxy Eicosatetraenoic Acid: number analyzed (Participants) | 36 | 36
  12-Hydroxy Eicosatetraenoic Acid | -0.00445 (0.491341) | -0.01181 (0.820744)
  15-Hydroxy Eicosapentaenoic Acid: number analyzed (Participants) | 8 | 12
  15-Hydroxy Eicosapentaenoic Acid | 0.00069 (0.025828) | 0.02028 (0.059147)
  19,20-diHydroxy Docosapentaenoic Acid: number analyzed (Participants) | 37 | 38
  19,20-diHydroxy Docosapentaenoic Acid | 0.16447 (0.865788) | 0.06606 (0.568695)
  8-Hydroxy Eicosatetraenoic Acid: number analyzed (Participants) | 30 | 28
  8-Hydroxy Eicosatetraenoic Acid | -0.00744 (0.093498) | 0.01879 (0.088266)
  Thiobarbituric Acid Reactive Substances: number analyzed (Participants) | 49 | 57
  Thiobarbituric Acid Reactive Substances | -0.0504 (0.79940) | 0.0406 (1.19656)
  Nitrotyrosine (NT3): number analyzed (Participants) | 49 | 57
  Nitrotyrosine (NT3) | -1.57 (72.964) | 10.35 (146.824)

17. Other Pre Specified Outcome: The Change in Metabolipidomic Profile in Blood, the Systemic Markers of Inflammation in Blood, the FEV1, the Body Weight and Calculated BMI
Description: Only in patients who experience a pulmonary exacerbation requiring IV antibiotics, this was to be assessed prior to- and after receiving an IV antibiotic course.
Time Frame: From baseline to 28 weeks
Population: Only very few subjects got sampled pre- and post-pulmonary exacerbation, rendering this data anecdotic. No outcome measure is presented.
Arm/Group | LAU-7b | Placebo
Number analyzed (Participants) | 0 | 0

18. Other Pre Specified Outcome: The Change From Baseline of Systemic Bone Formation and Resorption Biomarkers
Description: This was assessed through blood sampling on 2 occasions during the trial at Baseline and Week 24.
Time Frame: Baseline and 24 weeks
Population: Absolute change from Baseline at Week 24. Intent to treat population (ITT)
Measure: Mean (Standard Deviation); unit: Change in ug/L
Arm/Group | LAU-7b | Placebo
Number analyzed (Participants) | 83 | 83
Change in ug/L
  Aminoterminal Propeptide | -5.0 (14.90) | -4.5 (16.97)
  C-Telopeptide | -0.012 (0.2092) | 0.015 (0.1857)
  Osteocalcin | -1.46 (6.181) | 0.57 (5.703)

19. Other Pre Specified Outcome: The Change From Baseline of Bone Mineral Density
Description: This was assessed through Lumbar spine bone mineral density measured on 2 occasions during the trial at Baseline and at Week 28 in a subset of sites and on a voluntary basis. Bone mineral density in g/cm2 is then normalized and expressed as a Z-score distribution according to age and gender. A Z-score of 0 represents the population mean for the age and gender category, a -1 value or +1 value means below or above the population mean bone mineral density for the age and gender category, but considered normal. A -2.5 value indicates secondary osteoporosis, a worse outcome.
Time Frame: Baseline and 28 weeks
Population: Absolute change from Baseline at Week 24. Intent to treat population (ITT) in subjects volunteering to undergo bone density measurement
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | LAU-7b | Placebo
Number analyzed (Participants) | 6 | 11
Z-score | -0.18 (0.69) | 0.09 (0.28)

ADVERSE EVENTS:
Time Frame: 28 weeks
Arm/Group | LAU-7b | Placebo
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/83
Serious Adverse Events (participants affected / at risk) | 20/83 | 15/83
Other Adverse Events (participants affected / at risk) | 80/83 | 79/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LAU-7b (N=83) | Placebo (N=83)
Loss of visual contrast sensitivity (Eye disorders) | 1 | 0
Distal intestinal obstruction syndrome (Gastrointestinal disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 15 | 10
Appendicitis (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Traumatic intracranial hemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LAU-7b (N=83) | Placebo (N=83)
Delayed dark adaptation (Eye disorders) | 22 | 4
Night blindness (Eye disorders) | 15 | 2
Delayed light adaptation (Eye disorders) | 10 | 2
Glare (Eye disorders) | 9 | 6
Visual impairment (Eye disorders) | 9 | 2
Xanthopsia (Eye disorders) | 7 | 0
Photophobia (Eye disorders) | 6 | 4
Diarrhea (Gastrointestinal disorders) | 11 | 6
Abdominal pain (Gastrointestinal disorders) | 8 | 7
Nausea (Gastrointestinal disorders) | 6 | 7
Fatigue (General disorders) | 10 | 7
Pyrexia (General disorders) | 6 | 4
Chest discomfort (General disorders) | 5 | 4
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 22 | 22
Upper respiratory tract infection (Infections and infestations) | 13 | 8
Nasopharyngitis (Infections and infestations) | 6 | 3
Glucose urine present (Investigations) | 6 | 2
Blood glucose increased (Investigations) | 4 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 3
Headache (Nervous system disorders) | 14 | 10
Insomnia (Psychiatric disorders) | 4 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 23 | 24
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 11 | 13
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 | 11
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 7 | 13
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 9
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Acne (Skin and subcutaneous tissue disorders) | 6 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 3
Rash (Skin and subcutaneous tissue disorders) | 4 | 8

LIMITATIONS AND CAVEATS:
The APPLAUD study started enrollment in November 2018 and was conducted through the COVID-19 pandemic and during market introduction of ETI (elexacaftor/tezacaftor/ivacaftor) in the participating countries. However, the study protocol and the statistical plan were amended to address the higher dropout rates caused by these two factors during the clinical trial and to allow enrolment of patients stabilized on ETI as their background CFTR modulator therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-07-31): https://cdn.clinicaltrials.gov/large-docs/88/NCT03265288/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-03): https://cdn.clinicaltrials.gov/large-docs/88/NCT03265288/SAP_001.pdf